CLINICAL TRIAL: NCT00589901
Title: Phase II Study of an All-Oral Combination of Capecitabine (X) and Cyclophosphamide (C) in Patients With Anthracycline- and Taxane-Pretreated Metastatic Breast Cancer
Brief Title: An All-Oral Combination of Capecitabine and Cyclophosphamide in Patients With Metastatic Breast Cancer (MBC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Base of drug clinical trials, Fudan University Cancer Hospital, Fudan University Cancer Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200507CX
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2008-04-18 (Estimated); Status verified 2008-04

CONDITIONS: Breast Cancer
Keywords: metastatic breast cancer; capecitabine; synergistic effect; chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): phase II trial of capecitabine and cyclophosphamide in the management of metastatic breast cancer
  Interventions: Drug: capecitabine and cyclophosphamide

INTERVENTIONS:
Drug: capecitabine and cyclophosphamide — capecitabine 1000 mg/m2 oral Bid d1-14
  cyclophosphamide 65 mg/m2 oral Qd d1-14
  Other Names: Xeloda

SUMMARY:
The primary objective of this study is to evaluate the time to progression. Secondary objectives are safety, OS and pharmacogenetic analysis. Sixty patients will be enrolled into this study.

DETAILED DESCRIPTION:
Xeloda (capecitabine) is converted to 5-fluorouracil by thymidine phosphorylase, and cyclophosphamide is capable of upregulating the expression of thymidine phosphorylase suggesting a synergistic effect.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer
* Anthracycline and taxane pretreated metastatic breast cancer
* Have not been previously treated with capecitabine
* ECOG performance status of ≤ 1
* Are female and ≥ 18 and ≤ 70 years of age
* Have at least one target lesion according to the RECIST criteria

Exclusion Criteria:

* Pregnant or lactating women
* ECOG ≥ 2
* Have been treated with capecitabine
* Evidence of CNS metastasis
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix or a contralateral breast cancer
* Abnormal laboratory values: hemoglobin < 8.0 g/dl, neutrophils < 1.5×10^9/L, platelets < 100×10^9/L, serum creatinine > upper limit of normal (ULN), serum bilirubin > ULN, ALT and AST > 5×ULN, AKP > 5×ULN
* Serious uncontrolled intercurrent infection
* Life expectancy of less than 3 months

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
TTP (first treatment of this regimen to disease progression) | every two cycles

SECONDARY OUTCOMES:
side effects | all cycles
pharmacogenetic analysis | collect blood samples before this therapy

CONTACTS AND LOCATIONS:
Overall Officials: Zhonghua Wang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Fumoleau P, Largillier R, Clippe C, Dieras V, Orfeuvre H, Lesimple T, Culine S, Audhuy B, Serin D, Cure H, Vuillemin E, Morere JF, Montestruc F, Mouri Z, Namer M. Multicentre, phase II study evaluating capecitabine monotherapy in patients with anthracycline- and taxane-pretreated metastatic breast cancer. Eur J Cancer. 2004 Mar;40(4):536-42. doi: 10.1016/j.ejca.2003.11.007. PMID 14962720
- [Background] Endo M, Shinbori N, Fukase Y, Sawada N, Ishikawa T, Ishitsuka H, Tanaka Y. Induction of thymidine phosphorylase expression and enhancement of efficacy of capecitabine or 5'-deoxy-5-fluorouridine by cyclophosphamide in mammary tumor models. Int J Cancer. 1999 Sep 24;83(1):127-34. doi: 10.1002/(sici)1097-0215(19990924)83:13.0.co;2-6. PMID 10449619
- [Derived] Wang Z, Lu J, Leaw S, Hong X, Wang J, Shao Z, Hu X. An all-oral combination of metronomic cyclophosphamide plus capecitabine in patients with anthracycline- and taxane-pretreated metastatic breast cancer: a phase II study. Cancer Chemother Pharmacol. 2012 Feb;69(2):515-22. doi: 10.1007/s00280-011-1728-3. Epub 2011 Aug 27. PMID 21874317